CLINICAL TRIAL: NCT03151226
Title: A Prospective, Observational, Double-blind (Black-Box) Study Evaluating Incidence, Severity and Predictive Factors of Respiratory Depression and Sleep Disorder Pattern During Postoperative Neuraxial Opioid Analgesia in OSA Screened Negative With BMI>=35 Kg/m2 Obstetric Patients After Cesarean Delivery Using Current Standard Intermittent Postoperative Monitoring Compared to Continuous Pulse Oximetry/Capnography
Brief Title: OSA Screen Negative With Spinal Duramorph
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulty and feasibility issues
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00033095
Record Dates: First submitted 2015-08-31; First posted 2017-05-12 (Actual); Results first posted 2018-03-08 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Depression
Keywords: obstructive sleep apnea screen negative; respiratory depression; cesarean section
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capnography monitoring (Other): single arm, all subjects receiving duramorph will receive capnography monitoring
  Interventions: Device: Capnography monitoring

INTERVENTIONS:
Device: Capnography monitoring — capnography and pulse oximetry will be initiated in the recovery room and worn for 12-24 hours post delivery
  Other Names: pulse oximetry

SUMMARY:
Non emergent scheduled cesarean sections will be consented to participate in this study of patients who have screened negative for obstructive sleep apnea and who are also BMI>/= 35 to have capnography monitoring postoperatively. The capnography and pulse oximetry will be initiated in the post anesthesia care unit and be worn for 12-24 hours after delivery. Data will be retrieved after that time period in a deidentified fashion. Medication usage will be reviewed as well as the standard of care information from the duramorph monitoring will be retrieved.

ELIGIBILITY:
Inclusion Criteria:

* OSA screen negative per hospital protocol
* age 18 or greater
* BMI>35
* consent to participate to wear capnography and pulse oximetry monitoring devices post delivery

Exclusion Criteria:

* Spanish speaking only
* under age 18
* contraindication to receiving drugs utilized in delivery anesthetic

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Pan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Novant Health Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capnography Monitoring
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — not wear device correctly | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capnography Monitoring
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression/Suppression
Description: defined by values obtained utilizing capnography and pulse oximetry
Time Frame: up to 24 hours
Population: the 2 subjects who wore device did not wear the device enough to be evaluable data
Arm/Group | Capnography Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Capnography Monitoring
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes